CLINICAL TRIAL: NCT02626325
Title: Effect of High-carbohydrate or High-monounsaturated Fatty Acids on Blood Pressure: a Meta-analysis of Randomized Clinical Trials
Brief Title: Effect of High-carbohydrate or High-monounsaturated Fat on Blood Pressure: Meta-analysis of Randomized Clinical Trials
Acronym: CHO-MUFA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: CHO-MUFA Meta
Record Dates: First submitted 2015-12-07; First posted 2015-12-10 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Blood Pressure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: High-carbohydrate or High-monounsaturated fat diets

SUMMARY:
High saturated fat acids diets are associated with elevated blood pressure which is associated with cardiovascular morbidity and mortality. For this reason, a change of diet is recommended to manage blood pressure and prevent cardiovascular complications. To achieve this nutritional goal, a high-carbohydrate diet or high-monounsaturated fat diet can be advised in the replacement of a saturated fat diet.

Previous meta-analysis of Garg (1998) cited randomized articles with inconsistent blood pressure lowering after consumption of a high-monounsaturated-fat diet compared with a high-carbohydrate diet only in type 2 diabetes patients. Moreover, another meta-analysis of Shah et al. (2007) showed slightly high blood pressure on diets rich in carbohydrates than diets rich in cis-monounsaturated fat after randomized and nonrandomized articles.

For this reason, a new meta-analysis of a randomized clinical trial will be performed to clarify the effects of high-carbohydrate or high-monounsaturated fat diets on blood pressure. Results from this meta-analysis will help health professionals take important decisions on patient diet and minimize cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials
* Parallel or Crossover Design
* Duration: at least 3 weeks
* Isocaloric diet

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy and unhealthy (T2DM, hyperlipidemic, hypertensive)
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 3 weeks
Mean arterial pressure | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto; Elena Jovanovskie, MSc, Principal Investigator — Unity Health Toronto; Any de Castro Ruiz Marques, MSc, Study Director — Unity Health Toronto
Locations (1):
- Vladimir Vuksan, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Jovanovski E, de Castro Ruiz Marques A, Li D, Ho HVT, Blanco Mejia S, Sievenpiper JL, Zurbau A, Komishon A, Duvnjak L, Bazotte RB, Vuksan V. Effect of high-carbohydrate or high-monounsaturated fatty acid diets on blood pressure: a systematic review and meta-analysis of randomized controlled trials. Nutr Rev. 2019 Jan 1;77(1):19-31. doi: 10.1093/nutrit/nuy040. PMID 30165599